CLINICAL TRIAL: NCT06633146
Title: Outpatient Stroke Rehabilitation Supported by Nature Interventions
Brief Title: Stroke Rehabilitation Utilizing Therapeutical Methods Designed for Nature Environments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: University of Helsinki (Other); University of Jyvaskyla (Other); Tampere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HA/2233 Q062
Record Dates: First submitted 2024-07-03; First posted 2024-10-09 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Stress, Psychological; Post Traumatic Stress Disorder; Depression, Anxiety; Loneliness
Keywords: stroke; rehabilitation; social support; cognitive functions; activity
MeSH Terms: conditions — Stroke; Stress, Psychological; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: randomised controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nature intervention group (Experimental): Participants take part in therapeutic individual and group sessions organised in nearby nature by the research worker.
  Interventions: Behavioral: Therapies in nature
- Control group (No Intervention): Participants do not participate in organised sessions but are encouraged to maintain physical activity and social life.

INTERVENTIONS:
Behavioral: Therapies in nature — Therapeutic tasks in nature specifically designed for the study
  Arms: Nature intervention group

SUMMARY:
Outpatient participants with a recent stroke diagnoses receive complimentary rehabilitation. The nature interventions include ergo- and physiotherapeutic and neurocognitive tasks with the support of an psychotherapeutic frame designed to be performed in a nature environment.

DETAILED DESCRIPTION:
Patients with an acute stroke are recruited to the study when signing out from the acute hospital care services. The patients are selected randomly into two groups: intervention and control groups in proportions 1:1. During the four-week study period the partipants in the control group are encouraged to maintain light physical activity 1 to 3 times per week with or without company. The research worker contacts the participants every week. In the nature group the research worker organises individual nature visits in the nearby nature twice a week and encourages the participants to go outdoors with a close-one once a week. All interventional contacts in the nature group are performed in a ecopsychotherapeutical frame consisting of ergo- and physiotherapeutic and neurocognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke

Exclusion Criteria:

* Traumatic intracranial bleeding without stroke
* A malign, aggressive disease
* Severe aphasia or incapable of independent decision making

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The effect of nature interventions on PROMIS questionnaire | 4 weeks
  Self-assessed quality of life assessed by a PROMIS (patient-reported outcomes measurement information system) questionnaire. Time points measured wk 0 and wk 4, efficacy evaluated on the basis of the difference between these time points. An increase in the obtained score is considered a positive effect.

SECONDARY OUTCOMES:
The effect of nature interventions on moods assessed by GAD7 | 4 weeks
  Evaluation of anxiety scales by a GAD7 (generalised anxiety disorder 7) interview, the score of the questionnaire (0-21 points) is evaluated wk 0 and wk 4. A decrease in the total score is considered as a positive effect on moods.
The effect of nature-based intervention on neurocognitive functions in COMET questionnaire | 4 wk
  Assessment of the efficacy of nature-based neuropsychological tasks on neurocognitive functions by a cognitive test COMET (cognitive method) -questionnaire. The total score is evaluated wk0 and wk4. An increase in the total score is considered a positive effect.

OTHER OUTCOMES:
The effect of nature interventions on functional ability assessed by a validated questionnaire WHODAS | 4 weeks
  Self-assessed functional ability in everyday life with a validated questionnaire WHODAS (WHO disability assessment scale). The total scores are evaluated wk0 and wk4. An increase in the total score is considered a positive effect.
The effect of nature interventions on microbiome | 4 weeks
  Microbiological analyses from skin flake and stool samples
The effect of nature interventions on the activity of autonomic nervous system | 4 weeks
  The evaluation of the state of the autonomic nervous system by heart rate variability by a portable device.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Haveri, MD PhD, Principal Investigator — Wellbeing Services County of Paijat-Hame
Locations (1):
- Joint Authority for Päijät-Häme Social and Health Care, Lahti, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salonen K, Hyvonen K, Paakkolanvaara JV, Korpela K. Flow With Nature Treatment for Depression: Participants' Experiences. Front Psychol. 2022 Jan 5;12:768372. doi: 10.3389/fpsyg.2021.768372. eCollection 2021. PMID 35069344